CLINICAL TRIAL: NCT00453297
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Dose, Oral, Dose Escalation Phase 1 Study to Evaluate the Safety and Tolerance of MF 101 as Well as the Pharmacokinetics of Its Key Active Components in Healthy Post-Menopausal Women.
Brief Title: Phase I Study to Evaluate the Safety and Efficacy of MF101 as Well as the Pharmacokinetics of Its Key Active Components
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bionovo (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MF-101-003
Expanded Access: Available
Record Dates: First submitted 2007-03-26; First posted 2007-03-28 (Estimated); Last update posted 2008-08-29 (Estimated); Status verified 2008-08

CONDITIONS: Healthy
Keywords: Bionovo; MF101; Herbs; The primary goal of this study is to identify the highest safe oral dose of MF101 that is well tolerated in humans.

INTERVENTIONS:
Drug: MF101

SUMMARY:
This Phase I trial in healthy, post-menopausal women is designed as a double-blind, placebo-controlled, randomized, ascending single-dose safety trial. MF101 will be administered as a single oral dose to a total of 32 enrolled subjects between the ages of 40-65 years. Eight subjects will be assigned to each of four cohorts. Within each cohort, six subjects will be randomized to receive MF101 and two subjects will receive placebo. MF101 doses will be incrementally escalated until the stopping criteria are reached. If stopping criteria are reached before the fourth cohort receives dosing, the next cohort may receive a dose between the dose that was administered to the cohort exhibiting symptoms of MF101 toxicity and the next lower dose group.

DETAILED DESCRIPTION:
The primary goal of this study is to identify the highest safe oral dose of MF101 that is well tolerated in humans.

Secondary goals include: characterizing clinical symptoms of MF101 toxicity in healthy subjects and evaluating the dose-dependent pharmacokinetics of key MF101 active components after a single oral dose.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal females, in good health and between 40 and 65 years of age.
* Normal body mass index equal or greater than 18 but not greater than 36
* Postmenopausal as defined by 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 30 mlU/ml or 6 weeks post-surgical bilateral oophorectomy with or without hysterectomy, or hysterectomy with FSH levels > 30 mlU/ml.
* Ability to comprehend and a willingness to sign an informed consent form.
* Ability and willingness to understand and follow study procedures.
* Clinical laboratory evaluations within the reference range for the testing laboratory, unless regarded not clinically significant by the Principle Investigator.
* Must have had mammogram within the last 9 months.
* Negative urine test for selected drugs of abuse at screening and after check-in at the study unit.
* Negative hepatitis panel (including HBsAg and anti-HCV), and HIV antibody screens.
* No chronic medications being taken.
* Must have a primary care physician.

Exclusion Criteria:

* History or clinical manifestations of significant metabolic, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, hepatic, gall bladder, renal, urological, or psychiatric disorders.
* Dyslipidemia
* History of abnormal renal function, uncontrolled hypertension, or malignancies.
* History of breast, uterine or ovarian cancer or melanoma.
* History of brain aneurism or ischemic events.
* Febrile disease
* Autoimmune disorders such as lupus erythematosis, multiple sclerosis or rheumatoid arthritis.
* Severe vasomotor symptoms defined as > 7/day or >50/week.
* Abnormal mammogram or breast examination within the last 9 months suggestive of cancer.
* Abnormal Pap smear or pelvic examination within the last 9 months suggestive of cancer.
* Double-wall endometrial thickness that exceeds 5 mm measured on transvaginal ultrasound.
* Unexplained abnormal uterine bleeding within six months of enrollment.
* Pregnancy or lactating.
* History of deep vein thrombosis or pulmonary embolism requiring anticoagulation.
* History of hypersensitivity or allergies to any drug compound, including the constituents of MF101 unless approved by the Principle Investigator.
* History or presence of a clinically significant abnormal ECG (QTcB > 450msec at screening or variation in QTcB > 30msec at screening).
* Likely to need medication during the study including contraceptives.
* History of alcoholism or drug addiction within 1 year prior to study entry (i.e., prior to check-in on Day-1).
* Use of any tobacco products (including cigarette, pipe, cigar, chewing, nicotine patch, or nicotine gum) within 6 months prior to study entry.
* Receipt of any investigational drug within 60 days prior to study entry.
* Use of prescription medications known to possibly be effective for the treatment of hot flashes within three months of enrollment for oral or transdermal drugs, or within 6 months of enrollment for implanted or injected drugs.
* Use of raloxifene, tamoxifen or aromatase inhibitors within three months of enrollment.
* Use of any other prescription medication or any alcohol-containing products/medications within 14 days prior to study entry.
* Use of over-the-counter, non-prescription preparations, within 7 days prior to study entry.
* Use of any caffeine-containing products/medications within 72 hours prior to study entry.
* Donation of blood within 6 weeks prior to study entry or of plasma within 2 weeks prior to screening.
* Receipt of blood products within 2 months prior to study entry.
* Any other condition or prior therapy which, in the opinion of the Investigator, would make the subject unsuitable for this study.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2006-10; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Identify the highest oral dose of MF101 that is safe and tolerated in humans.
Number and type of adverse events
Clinical laboratory including: Chemistry, hematology, blood coagulation and urinalysis
Physical exam and vital signs

SECONDARY OUTCOMES:
Characterize MF101 toxicity and associated clinical symptoms in healthy subjects.
Establish cardiac safety (QTcB).
Study the dose dependent pharmacokinetics of MF101's key active components after oral administration.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Henthorn, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Health Sciences Center, Aurora, Colorado, United States